CLINICAL TRIAL: NCT05309057
Title: Effect of Intermittent Fasting Strategies on Cardiometabolic Risk: A Systematic Review and Network Meta-analysis of Randomized Controlled Trials
Brief Title: Network Meta-analysis of Intermittent Fasting and Cardiometabolic Risk
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, John Sievenpiper, Professor, University of Toronto
Other Study IDs: DNSG-IF
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Obesity; PreDiabetes; Diabetes; Hypertension; NAFLD; Metabolic Syndrome; Dyslipidemias; Inflammation; Gout; Cardiometabolic Syndrome; Cardiovascular Diseases
Keywords: Intermittent fasting; Continuous energy restriction; Weight loss; Systematic review and meta-analysis; Network metanalysis; Randomized controlled trial; Clinical practice guideline; Adiposity; Glycemic control; Blood pressure; Blood lipids; NAFLD markers; Uric acid; inflammatory markers; Cardiometabolic risk factors
MeSH Terms: conditions — Obesity; Prediabetic State; Diabetes Mellitus; Hypertension; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Dyslipidemias; Inflammation; Gout; Cardiovascular Diseases; Intermittent Fasting; Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Studies with intermittent fasting: Studies with intermittent fasting strategies.
  Interventions: Dietary Supplement: Intermittent Fasting

INTERVENTIONS:
Dietary Supplement: Intermittent Fasting — Methods of intermittent fasting strategies, continuous energy restriction, and ad libitum diet.

SUMMARY:
Intermittent fasting is a method of restricting calories over a defined period of time and includes regimens such as whole-day fasting, alternate-day fasting, and time-restricted feeding. There is emerging evidence that intermittent fasting or energy restriction might be more beneficial than continuous energy restriction for some risk factors. The effect of intermittent fasting on risk factors associated with obesity, diabetes, and cardiovascular disease, however, is not clear. The European Association for the Study of Diabetes (EASD) has yet to make any recommendations regarding the role of intermittent fasting in the management of diabetes. To inform the update of the EASD Clinical Practice Guidelines for Nutrition Therapy, tthe Diabetes and Nutrition Study Group (DNSG) of the EASD has commissioned a systematic review and network meta-analysis of randomized controlled trials of the effect of different intermittent fasting strategies on established cardiometabolic risk factors. The findings generated by this proposed knowledge synthesis will shape guide current guidelines and improve health outcomes by educating healthcare providers and patients, and by guiding future research design.

DETAILED DESCRIPTION:
Background: 'Intermittent fasting' is currently the most popular trending diet, yet its clinical utility remains unclear. Previous systematic reviews and meta-analyses of intermittent fasting have been limited by a narrow focus on weight loss, one specific method of intermittent fasting, and/or a subset of participants who would be the least likely to benefit. Other issues have included unexplained heterogeneity, incorrect analyses and/or lack of assessment of the certainty of the evidence. There is emerging evidence that intermittent fasting may improve cardiometabolic risk markers independent of calories. However, there is a lack of certainty about the effectiveness of intermittent fasting on overall cardiometabolic risk across different health conditions, and the differences between the various methods of intermittent fasting. The European Association for the Study of Diabetes (EASD) has yet to make any recommendations regarding the role of intermittent fasting in the management of diabetes. To inform the update of the EASD Clinical Practice Guidelines for Nutrition Therapy, the Diabetes and Nutrition Study Group (DNSG) of the EASD has commissioned a systematic review and network meta-analysis (an approach which has the advantage over traditional pairwise meta-analyses of being able to assess simultaneously multiple interventions) to assess the effect of the different strategies of intermittent energy restriction (intermittent fasting) versus continuous energy restriction and ad libitum diets on cardiometabolic risk in randomized controlled trials and assess the certainty of evidence using the Grading of Recommendations Assessment, Development and Evaluation (GRADE) approach.

Objective: To assess simultaneously the effect of the various strategies of intermittent energy restriction (intermittent fasting), continuous energy restriction, and ad libitum diets on body weight and other cardiometabolic risk factors in a systematic review and network meta-analysis of randomized trials using the GRADE approach.

Design: Each systematic review and meta-analysis will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses extension for network meta-analyses (PRISMA-Network).

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms. These searches will be supplemented by hand searches of references of included studies. Abstracts will be included and no language restrictions will be used.

Study selection: The investigators will include randomized controlled trials (RCTs) that are >=3-weeks duration investigating the effect of intermittent fasting, continuous caloric restriction and/or ad libitum diets on cardiometabolic risk factors in adults.

Data extraction: Two or more investigators will independently extract relevant data. Standard computations and imputations will be used to derive missing variance data. All disagreements will be resolved by consensus.

Risk of bias: Risk of bias will be assessed using the Cochrane Risk of Bias (RoB) Tool by the two or more investigators.

Outcomes: There will be 10 outcome clusters. The primary outcome will be body weight. Secondary outcomes will be other markers of adiposity (BMI, body fat, waist circumference); glycemic control (glycated blood proteins [HbA1c, fasting blood glucose, postprandial blood glucose, fasting blood insulin, homeostasis model assessment of insulin resistance [HOMA-IR]); established therapeutic lipid targets (LDL-cholesterol, non-HDL-cholesterol, apolipoprotein B [apo B], HDL-cholesterol, triglycerides); blood pressure (systolic blood pressure and diastolic blood pressure); markers of NAFLD (intrahepatocellular lipids [IHCL], alanine aminotransferase [ALT], aspartate aminotransferase [AST]); uric acid; and markers of inflammation (CRP).

Data synthesis: The investigators will perform a network meta-analysis comparing all the interventions simultaneously. These interventions will include alternate day fasting, cyclical whole day fasting, time restricted feeding, continuous energy restriction, and ad libitum diet in a single analysis by combining both direct and indirect evidence across the selected network of studies. Separate pooled analyses will be conducted for each cardiometabolic risk factor using the random-effects network meta-analysis. Intrasitivity will be adjudged using incoherence. Global method of incoherence (design-by-treatment interaction) and inconsistency factors (disagreement between direct and indirect estimates) will be used to estimate incoherence. A-priori subgroup analyses (health status, age, control diet energy restriction, diet supervision, study design, follow-up, feeding control, randomization, energy balance, baseline body weight, funding source, and ROB) will be performed. Separate analysis will be performed in people with diabetes. Publication bias will be assessed if there are ≥10 comparisons. The overall certainty of the evidence for each outcome will be assessed with GRADE using the CINeMA approach.

Evidence Assessment: The certainty of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE) approach.

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant decision makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed project will be the most comprehensive synthesis and evaluation of the totality of evidence on the role of intermittent fasting in cardiometabolic health. These findings will aid in strengthening current guidelines and improve health outcomes by informing shared clinical decision making between healthcare providers and patients and guiding future research.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled trials in humans
* Intermittent fasting intervention
* Continuous energy restriction, ad libitum diet, or other intermittent fasting diet as comparators
* Diet duration ≥1 weeks
* Data for at least one prespecified outcome
* Viable outcome data

Exclusion Criteria:

* Non-human studies
* Observational studies
* Children
* Multi-modal interventions
* Diet duration < 1 weeks
* No viable outcome data
* Lack of suitable comparator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults of all health statuses.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Body weight | Through study completion, up to 20 years
  Body weight in kg

SECONDARY OUTCOMES:
Adiposity - BMI | Through study completion, up to 20 years
  Body mass index (BMI) in kg/m2
Adiposity - Waist circumference | Through study completion, up to 20 years
  Waist circumference in cm
Adiposity - Body fat | Through study completion, up to 20 years
  Body fat in % (relative units)
Glycemic control - HbA1c | Through study completion, up to 20 years
  Glycemic control - HbA1c
Glycemic control - fasting plasma glucose (FPG) | Through study completion, up to 20 years
  Fasting plasma glucose (FPG) in mmol/L
Glycemic control - 2h plasma glucose (2h-PG) | Through study completion, up to 20 years
  2h plasma glucose (2h-PG) during a 75g oral glucose tolerance test (OGTT) in mmol/L
Glycemic control - fasting plasma insulin (FPI) | Through study completion, up to 20 years
  Fasting plasma insulin (FPI) in pmol/L
Glycemic control - homeostasis model assessment of insulin resistance (HOMA-IR) | Through study completion, up to 20 years
  Homeostasis model assessment of insulin resistance (HOMA-IR)
Established blood lipid targets - LDL-cholesterol (LDL-C) | Through study completion, up to 20 years
  LDL-cholesterol (LDL-C) in mmol/L
Established blood lipid targets - non-HDL-cholesterol (non-HDL-C) | Through study completion, up to 20 years
  non-HDL-cholesterol (non-HDL-C) in mmol/L
Established blood lipid targets - apolipoprotein B (apo B) | Through study completion, up to 20 years
  Apolipoprotein B (apo B) in g/L
Established blood lipid targets - triglycerides | Through study completion, up to 20 years
  Triglycerides in mmol/L
Established blood lipid targets - HDL-cholesterol (HDL-C) | Through study completion, up to 20 years
  HDL-cholesterol (HDL-C) in mmol/L
Blood pressure - Systolic blood pressure (SBP) | Through study completion
  Systolic blood pressure (SBP) in mmHg
Blood pressure - diastolic blood pressure (DBP) | Through study completion, up to 20 years
  Diastolic blood pressure (DBP) in mmHg
Markers of non-alcoholic fatty liver disease (NAFLD) - Intrahepatocellular lipids (IHCL) | Through study completion, up to 20 years
  Intrahepatocellular lipids (IHCL) in % (relative units)
Markers of non-alcoholic fatty liver disease (NAFLD) - alanine transaminase (ALT) | Through study completion, up to 20 years
  Alanine transaminase (ALT) in U/L
Uric acid | Through study completion, up to 20 years
  Uric acid in mmol/L
Markers of inflammation - CRP | Through study completion, up to 20 years
  CRP in mg/dL

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario
  - Faculty of Medicine, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Semnani-Azad Z, Khan TA, Chiavaroli L, Chen V, Bhatt HA, Chen A, Chiang N, Oguntala J, Kabisch S, Lau DC, Wharton S, Sharma AM, Harris L, Leiter LA, Hill JO, Hu FB, Lean ME, Kahleova H, Rahelic D, Salas-Salvado J, Kendall CW, Sievenpiper JL. Intermittent fasting strategies and their effects on body weight and other cardiometabolic risk factors: systematic review and network meta-analysis of randomised clinical trials. BMJ. 2025 Jun 18;389:e082007. doi: 10.1136/bmj-2024-082007. PMID 40533200